CLINICAL TRIAL: NCT06504004
Title: Chronic Neck Pain: A Comprehensive Study of the Relationship Between Cognitive Function and Functional Status
Brief Title: Chronic Neck Pain and Cognitive Function
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Collaborators: Bozok University (Other)
Responsible Party: Principal Investigator, T Dere, Physiotherapist, Hacettepe University
Other Study IDs: YBozok
Record Dates: First submitted 2024-07-03; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Neck Pain; Cognitive Symptom
Keywords: Neck pain; cognitive function; functional status
MeSH Terms: conditions — Neck Pain; Neurobehavioral Manifestations

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: The aim of this study was to investigate the relationship between cognitive function and pain, functional limitations, and cervical muscle endurance in individuals with chronic neck pain (CNP).

Methods: The study included 29 individuals (28F, 1M) aged between 18 and 65 years, with non-specific neck pain lasting for at least 3 months, non-neurological symptoms, and no history of head, neck or upper extremity surgery in the last 6 months. Cognitive functions were assessed using the Montreal Cognitive Assessment (MOCA) and Trail Making Test (TMT), pain level using the Visual Analog Scale (VAS) and Bournemouth Neck Pain Questionnaire (BNPQ), functional limitations using the The Profile Fitness Mapping neck questionnaire (ProFitMap-neck) and muscle endurance using cervical flexor, extensor, and deep flexor muscle endurance tests.

DETAILED DESCRIPTION:
The study was conducted with ethical approval from the ________ University Ethics Committee (Approval number: 111/2023, Approval Date: 09/12/2023) to investigate the relationship between cognitive functions and functional status in individuals with chronic neck pain. The study adhered to the principles of the Declaration of Helsinki. Power analysis was performed using 'Correlation' with an effect size of 0.5 for the sample size. The statistical test employed in this study was the point biserial model, and the analysis type was 'A priori: Compute required sample size' using G*Power 3.1.9.2 version (Heinrich-Heine-Universität in Düsseldorf, Germany). For the post-hoc power analysis test, the r value between functional limitations and TMT-A test scores was used. It was determined that the study had 90% power with 29 participants.

It is worth noting that all individuals participating in the study provided written informed consent. The study involved individuals between the ages of 18 and 65 who had been experiencing neck pain at rest with a score of 3 or more on the VAS for at least 3 months. It was ensured that these individuals did not have any neurological deficits or pathological findings, such as fracture, dislocation, tumor, or infection, in radiological examinations. Exclusion criteria for the study included individuals with neurological or psychiatric diseases, a history of head trauma resulting in loss of consciousness, epilepsy, a history of neurosurgical intervention, intracranial hypertension, cancer, diabetes, dementia, brain dysfunction, psychological problems such as depression and anxiety diagnosed by a specialist physician and receiving treatment for these diseases, as well as individuals who were illiterate.

Assessment of Pain Severity The study evaluated the degree of neck pain experienced by individuals with chronic neck pain using two different methods: the 10 cm Visual Analogue Scale (VAS) developed by Price et al. Price et al. 1983) and the Bournemouth Neck Pain Questionnaire (BNPQ) developed by Bolton et al (Bolton & Humphreys 2002). Participants were asked to indicate their level of neck pain on a 10 cm horizontal line, where 0 indicates no pain and 10 indicates unbearable pain, during rest, at night, and during activity. BNPQ evaluates individuals with neck pain based on pain intensity, participation in family and social life, depression, anxiety, kinesiophobia, coping skills with pain in the last week, and other relevant factors. The questionnaire consists of 7 questions, and individuals are asked to score each question on a scale of 0 to 10. The total score ranges from 0 to 70, with higher scores indicating more severe neck pain. Telci et al. conducted a study to assess the validity and reliability of the questionnaire in the Turkish population.

Assessment of Cognitive Status The cognitive status of individuals with chronic neck pain was assessed in the study using the Montreal Cognitive Assessment (MoCA) and Trail Making Test (TMT). The MoCA, a tool for detecting mild cognitive impairment, was developed by Nasreddine et al (Nasreddine et al. 2005). Its Turkish validity and reliability were established by Selekler et al. The total score ranges from 0 to 30, with a score of 26 and above indicating normal cognitive status. TMT is a cognitive assessment tool that evaluates various cognitive functions, including visual-motor coordination, conceptual scanning, motor speed, planning, numerical knowledge, abstract thinking, tendency to react based on the physical characteristics of the stimulus, set switching, concentration, and movement. The questionnaire is divided into two parts, Part A and Part B. Part A assesses psychomotor speed and attention, while Part B assesses executive functions such as set switching, visual scanning speed, and visual alertness. Turkish validity and reliability of the questionnaire was performed by Türkeş et al. (Türkeş et al. 2015).

Evaluation of Functional Status The Profit Neck Mapping Questionnaire (ProFitMap-Neck) was implemented to assess the symptoms and functional limitations of individuals with chronic neck pain. The questionnaire consists of 26 items, including pain, tension, sensation, and balance, which are scored for frequency and severity of each symptom, resulting in two separate scores: symptom frequency score and symptom severity score. The functional limitation scale assesses the difficulty of performing activities such as lifting weights and wearing a t-shirt, resulting in a functional limitation score ranging from 0-100. An increase in the score indicates an improvement in functional status (Björklund et al. 2012).

Stabilizer biofeedback was used to evaluate the endurance of the deep cervical flexor muscles. Patients in a supine position had the stabilizer placed on their cervical region and were instructed to slowly nod their head, simulating a 'yes' movement. The test ranged from 20 mmHg to 30 mmHg, with the pressure needing to be sustained for 10 seconds at every 2 mmHg increase without interruption. The activation score and performance index were determined by evaluating the patient's capacity to execute and sustain 10 repetitions over a 10-second interval at a particular pressure level. The activation score had a maximum value of 10 mmHg, whereas the performance index had a maximum value of 100 (Jull, O'Leary & Falla 2008). To evaluate the endurance of the neck extensor muscles, a 2 kg weight was attached to the participants at the C6 level using a 10 cm band while lying prone. The maximum time they could maintain an upright head position was measured in seconds (Andias, Neto & Silva 2018) and recorded. Additionally, the endurance of the cervical flexor muscles was assessed using the cervical flexor muscle endurance test. According to this test, the maximum time that an individual could lift and hold their head at a height of approximately 2.5 cm in a supine hooked position with their hands on their abdomen and chin retracted was recorded (Domenech et al. 2011).

Statistical analysis The descriptive statistics of continuous variables were presented as the mean and standard deviation or the median and quartile, in accordance with the normality assumption. For categorical variables, the frequency (%) was given. All reported p-values were two-tailed. The data were analysed using IBM SPSS Statistics for Windows v.23.0. An examination was conducted to ascertain whether the assumption of normal distribution for the data was satisfied. The results supported the use of the Pearson correlation coefficient, with the exception of certain variables, for which the Spearman correlation coefficient was employed. A significance level of p < 0.05 was established (Fitzgerald etal. 2004).

ELIGIBILITY:
Inclusion Criteria:

* It is worth noting that all individuals participating in the study provided written informed consent. The study involved individuals between the ages of 18 and 65 who had been experiencing neck pain at rest with a score of 3 or more on the VAS for at least 3 months.

Exclusion Criteria:

* It was ensured that these individuals did not have any neurological deficits or pathological findings, such as fracture, dislocation, tumor, or infection, in radiological examinations.
* Neurological or psychiatric diseases, a history of head trauma resulting in loss of consciousness, epilepsy, a history of neurosurgical intervention, intracranial hypertension, cancer, diabetes, dementia, brain dysfunction, psychological problems such as depression and anxiety diagnosed by a specialist physician and receiving treatment for these diseases
* Individuals who were illiterate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: It is worth noting that all individuals participating in the study provided written informed consent. The study involved individuals between the ages of 18 and 65 who had been experiencing neck pain at rest with a score of 3 or more on the VAS for at least 3 months.
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Pain-Visual Analogue Scale (VAS) | Jun 2024
  The study evaluated the degree of neck pain experienced by individuals with chronic neck pain using two different methods: the 10 cm Visual Analogue Scale (VAS) developed by Price et al. Price et al. 1983). Participants were asked to indicate their level of neck pain on a 10 cm horizontal line, where 0 indicates no pain and 10 indicates unbearable pain, during rest, at night, and during activity
Pain-Bournemouth Neck Pain Questionnaire (BNPQ) | Jun 2024
  BNPQ evaluates individuals with neck pain based on pain intensity, participation in family and social life, depression, anxiety, kinesiophobia, coping skills with pain in the last week, and other relevant factors. The questionnaire consists of 7 questions, and individuals are asked to score each question on a scale of 0 to 10. The total score ranges from 0 to 70, with higher scores indicating more severe neck pain. Telci et al. conducted a study to assess the validity and reliability of the questionnaire in the Turkish population.
Assessment of Cognitive Status-Montreal Cognitive Assessment (MoCA) | Jun 2024
  The MoCA, a tool for detecting mild cognitive impairment, was developed by Nasreddine et al (Nasreddine et al. 2005). Its Turkish validity and reliability were established by Selekler et al. The total score ranges from 0 to 30, with a score of 26 and above indicating normal cognitive status.
Assessment of Cognitive Status-Trail Making Test (TMT) | Jun 2024
  TMT is a cognitive assessment tool that evaluates various cognitive functions, including visual-motor coordination, conceptual scanning, motor speed, planning, numerical knowledge, abstract thinking, tendency to react based on the physical characteristics of the stimulus, set switching, concentration, and movement. The questionnaire is divided into two parts, Part A and Part B. Part A assesses psychomotor speed and attention, while Part B assesses executive functions such as set switching, visual scanning speed, and visual alertness. Turkish validity and reliability of the questionnaire was performed by Türkeş et al. (Türkeş et al. 2015).
Evaluation of Functional Status-Profit Neck Mapping Questionnaire (ProFitMap-Neck) | Jun 2024
  The Profit Neck Mapping Questionnaire (ProFitMap-Neck) was implemented to assess the symptoms and functional limitations of individuals with chronic neck pain. The questionnaire consists of 26 items, including pain, tension, sensation, and balance, which are scored for frequency and severity of each symptom, resulting in two separate scores: symptom frequency score and symptom severity score. The functional limitation scale assesses the difficulty of performing activities such as lifting weights and wearing a t-shirt, resulting in a functional limitation score ranging from 0-100. An increase in the score indicates an improvement in functional status (Björklund et al. 2012).
Evaluation of Functional Status-Stabilizer biofeedback | Jun 2024
  Stabilizer biofeedback was used to evaluate the endurance of the deep cervical flexor muscles. Patients in a supine position had the stabilizer placed on their cervical region and were instructed to slowly nod their head, simulating a 'yes' movement. The test ranged from 20 mmHg to 30 mmHg, with the pressure needing to be sustained for 10 seconds at every 2 mmHg increase without interruption. The activation score and performance index were determined by evaluating the patient's capacity to execute and sustain 10 repetitions over a 10-second interval at a particular pressure level.
Evaluation of Functional Status-Cervical Flexor Endurance Test | Jun 2024
  the endurance of the cervical flexor muscles was assessed using the cervical flexor muscle endurance test. According to this test, the maximum time that an individual could lift and hold their head at a height of approximately 2.5 cm in a supine hooked position with their hands on their abdomen and chin retracted was recorded (Domenech et al. 2011).

CONTACTS AND LOCATIONS:
Overall Officials: Tuğba Dere, MSc, Principal Investigator — Yozgat Bozok University
Locations (1):
- School of Sarıkaya Physical Therapy and Rehabilitation, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Beltran-Alacreu H, Lopez-de-Uralde-Villanueva I, Calvo-Lobo C, Fernandez-Carnero J, La Touche R. Clinical features of patients with chronic non-specific neck pain per disability level: A novel observational study. Rev Assoc Med Bras (1992). 2018 Aug;64(8):700-709. doi: 10.1590/1806-9282.64.08.700. PMID 30673040
- [Background] Bjorklund M, Hamberg J, Heiden M, Barnekow-Bergkvist M. The ProFitMap-neck--reliability and validity of a questionnaire for measuring symptoms and functional limitations in neck pain. Disabil Rehabil. 2012;34(13):1096-107. doi: 10.3109/09638288.2011.635747. Epub 2011 Dec 12. PMID 22149067
- [Result] Hyland-Monks R, Cronin L, McNaughton L, Marchant D. The role of executive function in the self-regulation of endurance performance: A critical review. Prog Brain Res. 2018;240:353-370. doi: 10.1016/bs.pbr.2018.09.011. Epub 2018 Oct 17. PMID 30390840
- [Result] Zhao H, Alam A, Chen Q, A Eusman M, Pal A, Eguchi S, Wu L, Ma D. The role of microglia in the pathobiology of neuropathic pain development: what do we know? Br J Anaesth. 2017 Apr 1;118(4):504-516. doi: 10.1093/bja/aex006. PMID 28403399